CLINICAL TRIAL: NCT06120309
Title: New Prognostic Index for Neoadjuvant Chemotherapy Outcome in Patients With Advanced High-grade Serous Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-963-01
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer; Neoadjuvant Chemotherapy; Prognostic Cancer Model
Keywords: High-grade serous ovarian cancer; Neoadjuvant chemotherapy; Prognostic index
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NACT Group
  Interventions: Diagnostic Test: CRS scoring; Diagnostic Test: Routine blood laboratory testing before treatment

INTERVENTIONS:
Diagnostic Test: CRS scoring — For pathological evaluation, the omental specimens resected during the IDS were stained with haematoxylin and eosin (H&E) and reviewed independently by two gynecologic pathologists, both blinded to the clinical data and each other's results. The pathology slide obtained from omentum, usually the site with the most viable tumor, was selected for CRS assessment according to the three-tiered CRS system recommended by 2019 ESMO ovarian cancer guidelines
Diagnostic Test: Routine blood laboratory testing before treatment — The routine blood tests and tumor marker measurements, including CA125, HE4, and inflammation-related serum biomarkers including neutrophils, lymphocytes, monocytes, fibrinogen, and platelets, were conducted within three days before the first NACT.

SUMMARY:
A validated prognostic index for the outcome of advanced high-grade serous ovarian cancer (HGSOC) patients undergoing neoadjuvant chemotherapy (NACT) is still lacking. To address this need, we developed an ovarian neoadjuvant chemotherapy prognostic index (ONCPI) to improve predictive accuracy. We analyzed the clinicopathological characteristics of advanced HGSOC patients receiving platinum-based NACT. Blood inflammatory composite markers were calculated and binary-transformed using optimal cutoffs. Omental hematoxylin and eosin (H&E) stained slides were selected for the assessment of chemotherapy response score (CRS). Logistic regression analysis and Cox proportional hazards regression model were utilized to develop a prognostic index.

DETAILED DESCRIPTION:
1. The clinicopathological data of patients newly diagnosed with high-grade serous ovarian cancer in Sun Yat-sen Memorial Hospital were collected and screened.
2. Statistical analysis of hematological indicators that may be related to inflammation before platinum-based therapy in patients who met the inclusion criteria, including but not limited to: Absolute white blood cell count, absolute neutrophil count, absolute lymphocyte count, absolute monocyte count, platelet count, hemoglobin and fibrinogen were calculated. NLR, MLR, PLR, FLR and SII were calculated, and the correlation between the above indicators and tumor grade, stage, platinum-based drug sensitivity and prognosis was analyzed.
3. CRS scoring was performed using H&E sections of omentum obtained during IDS surgery.
4. logistic regression and Cox regression were used to analyze the independent risk factors affecting the sensitivity of neoadjuvant platinum-based chemotherapy and the prognosis of patients.
5. K-M analysis and ROC curve were used to analyze the predictive value of NLR combined with CRS ONCPI index for the response of high-grade serous ovarian cancer to platinum therapy.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of HGSOC by two experienced pathologists;
2. clinical stage III-IV according to the 2018 International Federation of Gynecology and Obstetrics (FIGO) guideline;
3. Eastern Cooperative Oncology Group (ECGO) performance status of 0 to 1;
4. no prior anti-cancer therapy;
5. received ≥ 3 cycles of platinum-based NACT followed by IDS;
6. complete pretreatment blood test results and clinical and imaging data.

Exclusion Criteria:

1. other pathological types;
2. without NACT or IDS;
3. incomplete pretreatment data;
4. lost to follow-up.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced HGSOC receiving platinum-based neoadjuvant chemotherapy (NACT) before interval debulking surgery (IDS) and postoperative adjuvant chemotherapy were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 465 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response to platinum-based chemotherapy | At least 6 months after initial chemotherapy
  After NACT-IDS and postoperative adjuvant chemotherapy, treatment efficacy was assessed according to NCCN guidelines. For primary tumor, patients who relapsed 6 months or more after initial chemotherapy were termed platinum-sensitive. In contrast, patients whose disease recurred in less than 6 months were classified as platinum-resistant.

SECONDARY OUTCOMES:
3-year progression-free survival (PFS) | 3 years
  PFS was calculated from the date of the first NACT until disease progression or death due to any cause.
3-year overall survival (OS) | 3 years
  OS was calculated from the date of the first NACT administration until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
If IPD is to be shared, it will be limited to the patient's clinicopathological and prognostic data, and the patient's personal information will be protected

REFERENCES:
- [Result] Hudry D, Becourt S, Scambia G, Fagotti A. Primary or Interval Debulking Surgery in Advanced Ovarian Cancer: a Personalized Decision-a Literature Review. Curr Oncol Rep. 2022 Dec;24(12):1661-1668. doi: 10.1007/s11912-022-01318-9. Epub 2022 Aug 15. PMID 35969358
- [Result] Colombo N, Sessa C, du Bois A, Ledermann J, McCluggage WG, McNeish I, Morice P, Pignata S, Ray-Coquard I, Vergote I, Baert T, Belaroussi I, Dashora A, Olbrecht S, Planchamp F, Querleu D; ESMO-ESGO Ovarian Cancer Consensus Conference Working Group. ESMO-ESGO consensus conference recommendations on ovarian cancer: pathology and molecular biology, early and advanced stages, borderline tumours and recurrent diseasedagger. Ann Oncol. 2019 May 1;30(5):672-705. doi: 10.1093/annonc/mdz062. PMID 31046081
- [Result] Liang WF, Wang LJ, Li H, Liu CH, Wu MF, Li J. The added value of CA125 normalization before interval debulking surgery to the chemotherapy response score for the prognostication of ovarian cancer patients receiving neoadjuvant chemotherapy for advanced disease. J Cancer. 2021 Jan 1;12(3):946-953. doi: 10.7150/jca.52711. eCollection 2021. PMID 33403051
- [Result] Li C, Wu J, Jiang L, Zhang L, Huang J, Tian Y, Zhao Y, Liu X, Xia L, E H, Gao P, Hou L, Yang M, Ma M, Su C, Zhang H, Chen H, She Y, Xie D, Luo Q, Chen C. The predictive value of inflammatory biomarkers for major pathological response in non-small cell lung cancer patients receiving neoadjuvant chemoimmunotherapy and its association with the immune-related tumor microenvironment: a multi-center study. Cancer Immunol Immunother. 2023 Mar;72(3):783-794. doi: 10.1007/s00262-022-03262-w. Epub 2022 Sep 3. PMID 36056951
- [Result] Rodolakis I, Pergialiotis V, Liontos M, Haidopoulos D, Loutradis D, Rodolakis A, Bamias A, Thomakos N. Chemotherapy Response Score in Ovarian Cancer Patients: An Overview of Its Clinical Utility. J Clin Med. 2023 Mar 10;12(6):2155. doi: 10.3390/jcm12062155. PMID 36983157